CLINICAL TRIAL: NCT02780739
Title: An Integrative System for Enhancing Fluid Intelligence (Gf) Through Human Cognitive Activity, Fitness, High-definition Transcranial Direct-current Brain Stimulation (HD-tDCS), and Nutritional Intervention
Brief Title: INSIGHT, A Comprehensive, Multidisciplinary Brain Training System
Acronym: INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: The City College of New York (Other); Aptima, Inc. (Unknown); Georgia Institute of Technology (Other); Circinnus LLC (Unknown); Autonomous University of Madrid, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2014-1312170004-Ph1a; 14212 (Other: UIllinoisUC IRB)
Record Dates: First submitted 2016-05-16; First posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Cognitive Ability, General
Keywords: Psychological Tests; Neuropsychological Tests; Transcranial Direct Current Stimulation; Exercise; Circuit-Based Exercise; Video Games; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Cognition; Executive Function; Learning; Problem Solving; Transfer (Psychology); Decision Making; Brain; Gray Matter; White Matter
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cognitive Training - 48 sessions (Experimental): 56 hours of video game training with Mind Frontiers adaptive cognitive training software (48 70-min sessions distributed over 16 weeks)
  Interventions: Behavioral: Cognitive Training - 48 sessions
- Fitness, Cognitive Training, sham tDCS (Experimental): 32 hours and 40 min of high-intensity cardiorespiratory fitness training (28 70-min sessions distributed over 16 weeks); 23 hours and 20 min of video game training with Mind Frontiers adaptive cognitive training software with simultaneous sham tDCS (20 70-min sessions distributed over weeks 5-16)
  Interventions: Behavioral: Fitness; Device: sham tDCS; Behavioral: Cognitive Training - 20 sessions
- Fitness, Cognitive Training, active tDCS (Experimental): 32 hours and 40 min of high-intensity cardiorespiratory fitness training (28 70-min sessions distributed over 16 weeks); 23 hours and 20 min of video game training with Mind Frontiers 1.0 adaptive cognitive training software with simultaneous active tDCS for a total of 10 hrs (20 70-min sessions distributed over weeks 5-16)
  Interventions: Behavioral: Fitness; Device: active tDCS; Behavioral: Cognitive Training - 20 sessions
- Active Control (Active Comparator): 56 hours of video game training with visual search and change detection tasks using open sesame software (48 70-min sessions distributed over 16 weeks)
  Interventions: Behavioral: Active Control
- No Contact Control (No Intervention): Completed no study activities for 16 weeks after pre-assessment, then returned for post-assessment

INTERVENTIONS:
Behavioral: Cognitive Training - 48 sessions — Mind Frontiers cognitive training software (Aptima Inc.) is a Wild West-themed Android application played on Nexus 10 tablets. This intervention includes 20 70-min sessions (23.33 hrs) completed over 12 weeks: 1/wk weeks 5-8, 2/wk weeks 9-16. The 6 mini-games, played in random order for 10 min each session, are Ante Up (Tower of London, executive functioning); Irrigator (visuospatial reasoning); Pen 'Em Up (dual task switching, executive function); Supply Run (Keep Track, working memory updating); Riding Shotgun (visuospatial working memory); and Sentry Duty (dual n-back, working memory). There is also a meta-game in which players build a town using resources earned from the mini-games, played for 5 min each session.
  Other Names: Mind Frontiers adaptive cognitive training - 48 sessions
  Arms: Cognitive Training - 48 sessions
Behavioral: Fitness — Based on high intensity cardiovascular resistance training (HICRT), this intervention includes a combination of aerobic and strength training. Sessions are conducted in a group of ≤20 participants per class, with ≤5 participants per trainer. This intervention includes 28 70-min sessions (32.67 hrs) completed over 16 weeks: 3/wk weeks 1-4, 2/wk weeks 5-8, 1/wk weeks 9-16. At the first and last session, participants complete the Army Physical Readiness Test. All other sessions consist of: Warm-up; Walk/Run; 2 HICRT circuits with 3 sets of 3-4 exercises; 1-2 min jump rope and 4-min power series between HICRT segments; Drills & Skills; and Cool-down/stretch.
  Other Names: high intensity cardiovascular resistance training; aerobic and strength training
  Arms: Fitness, Cognitive Training, active tDCS; Fitness, Cognitive Training, sham tDCS
Behavioral: Active Control — The active control condition consists of 2 tasks (change detection and visual search) with 3 variants each. This intervention includes 48 70-min sessions (56 hrs) completed over 16 weeks: 3/wk. The 6 tasks are played in random order for 10 min each session.
  Other Names: Adaptive Visual Search/Change Detection
  Arms: Active Control
Device: active tDCS — Active HD-tDCS is administered during the first 30 minutes of each Mind Frontiers session. Therefore, the schedule is 20 30-min sessions (10 hrs) completed over 12 weeks: 1/wk weeks 5-8, 2/wk weeks 9-16. The HD-tDCS devices are Soterix Medical 2x2 models, using 4 electrodes (2 anodal and 2 cathodal). Electrodes are held in place with custom, 3D-printed electrode holders inserted into EEG caps, using EEG gel. Participants receive 2.0 mA current for 30 min, split over the 2 anodal electrodes, each drawing ≤1.0 mA. Stimulation is ramped up and ramped down over 30 sec at the beginning and end of the 30-min stimulation period.
  Other Names: active high-def transcranial direct current stimulation
  Arms: Fitness, Cognitive Training, active tDCS
Device: sham tDCS — Sham HD-tDCS is administered during the first 30 minutes of each Mind Frontiers session. Therefore, the schedule is 20 30-min sessions (10 hrs) completed over 12 weeks: 1/wk weeks 5-8, 2/wk weeks 9-16. The HD-tDCS devices are Soterix Medical 2x2 models, using 4 electrodes (2 anodal and 2 cathodal). Electrodes are held in place with custom, 3D-printed electrode holders inserted into EEG caps, using EEG gel. Participants do not receive sustained stimulation; it is ramped up and ramped down over 30 sec at the beginning and end of the 30-min stimulation period to elicit the sensation of simulation and make the sham condition more convincing.
  Other Names: sham high-definition transcranial direct current stimulation
  Arms: Fitness, Cognitive Training, sham tDCS
Behavioral: Cognitive Training - 20 sessions — Mind Frontiers cognitive training software (Aptima Inc.) is a Wild West-themed Android application played on Nexus 10 tablets. This intervention includes 20 70-min sessions (23.33 hrs) completed over 12 weeks: 1/wk weeks 5-8, 2/wk weeks 9-16. The 6 mini-games, played in random order for 10 min each session, are Ante Up (Tower of London, executive functioning); Irrigator (visuospatial reasoning); Pen 'Em Up (dual task switching, executive function); Supply Run (Keep Track, working memory updating); Riding Shotgun (visuospatial working memory); and Sentry Duty (dual n-back, working memory). There is also a meta-game in which players build a town using resources earned from the mini-games, played for 5 min each session.
  Other Names: Mind Frontiers adaptive cognitive training - 20 sessions
  Arms: Fitness, Cognitive Training, active tDCS; Fitness, Cognitive Training, sham tDCS

SUMMARY:
Adaptive reasoning and problem-solving are critical skills that allow for accurate decisions to be made based on varying levels of information. In many situations these decisions must be made and communicated under stressful, time-sensitive conditions. In such contexts, an ability to apply inductive and deductive reasoning to complex, ambiguous, and/or novel problems is critical. The objective of the INSIGHT project is to establish a comprehensive and rigorous brain training protocol to significantly improve adaptive reasoning and problem solving. We will examine a variety of interventions (cognitive training, physical fitness training, physiological stimulation, , and combinations thereof) to assess their ability to improve adaptive reasoning and problem solving abilities. Multimodal interventions are hypothesized to act synergistically to significantly enhance fluid intelligence (Gf) and underlying brain structure and function.

DETAILED DESCRIPTION:
Recent innovations in cognitive neuroscience have advanced understanding of the neurobiological foundations of fluid intelligence (Gf) and adaptive reasoning and problem solving (ARP). Rather than engaging a single brain structure (e.g., prefrontal cortex) or operating at a fixed level of performance throughout adulthood, emerging neuroscience evidence indicates that Gf and ARP are mediated by a distributed neural system whose functions can be significantly enhanced by specific types of interventions, including cognitive training, high-definition transcranial direct-current brain stimulation (HD-tDCS), and physical fitness training. The main objective of the INSIGHT project is to establish and validate a comprehensive and rigorous brain training protocol that incorporates the best available interventions for the enhancement of Gf and ARP.

The project was divided into two phases, with the first occurring in February -November 2014 and the second occurring February - December 2015. The two phases were similar in structure and goals/hypotheses, but had several methodological differences in terms of interventions, arms, and outcome measures. This document contains information pertinent to only the 2014 phase, which examined the relative contributions of physical fitness intervention, video-game based training, and high-definition transcranial direct-current brain stimulation (HD-tDCS) to the improvement of Gf/ARP, executive function, working memory, relational memory, physical fitness level, and brain structure/function.

Arms/groups completed 1 week of testing to establish baseline measurements of cognitive abilities, physical fitness, and brain structure/function. 16 weeks of various intervention protocols. These protocols could include single or multiple intervention type(s) with varying schedules. Three 70-min training sessions were completed per week, so all arms completed 56 hours of training, total. Following completion of the intervention period was 1 week of post-assessment to measure changes in cognitive abilities, physical fitness, and brain structure/function.

Technical Justification for Physical Fitness Intervention: The beneficial effects of physical fitness on cognitive performance and brain health have been documented in many studies. For example, this literature suggests that increased exercise leads to the birth of new neurons in the hippocampus (a key brain region underlying Gf), increased connections among neurons throughout the brain, the development of new vasculature structure, increased production of neurotrophic proteins, enhanced learning and memory, and enhanced executive control including attention and inhibition, working memory, mental flexibility, and action monitoring. In particular, (1) exercise effects are largest for tasks that involve executive control functions for working memory, planning, and problem solving - abilities that are essential for Gf and ARP; and (2) aerobic exercise training, when combined with strength and flexibility training, had a greater positive effect on cognition compared to exercise training programs that included only aerobic components. Such findings provide important justification for the physical activity intervention proposed here. Hence, the proposed fitness intervention employs a combined aerobic/resistance training program to further enhance the benefits of cognitive training on Gf and ARP.

Technical Justification for Video Game-Based Training: Training on five cognitive skills - (1) processing speed, (2) attention, (3) working memory, (4) relational memory, and (5) cognitive flexibility - has been shown to provide promising transfer results to Gf and other relevant constructs. This training regime is the basis for the design of the Mind Frontiers software platform. Mind Frontiers includes an integrated suite of mini-games that are designed to train these five core cognitive skills. The mechanics, as abstractions of the cognitive exercises, ensure that the scientific integrity and the training effect of the exercises are preserved, but the exercises are implemented as games with motivational features and adaptive difficulty.

Technical justification for HD-tDCS: It has been hypothesized that Gf and ARP are critically dependent on a fronto-parietal brain network, and thus that bilateral, specific stimulation of the frontal cortex with high definition transcranial direct current stimulation (HD-tDCS) would have an excitatory effect on neurons within that network, making them more likely to fire, and thereby enabling faster learning and facilitating transfer to Gf.

Technical Justification for Active Control: Change detection and visual search tasks were selected as the active control tasks because previous work had indicated that training low-level perceptual abilities did not transfer to Gf and ARP.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* US citizen, US permanent resident, or student/work visa sponsored by UIUC
* Available for 18-20 weeks
* Ages 18 - 44
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing

Exclusion Criteria:

* Previous participant in studies with similar protocols
* Currently taking any medication affecting CNS
* Has taken medication affecting CNS in past 2 months
* Current or planned pregnancy
* Recurrent migraines
* Concussion in past 2 years
* History of stroke
* History of epilepsy/seizures
* Any medical condition affecting CNS (e.g., history of thyroid cancer)
* Any medical condition affecting capability to exercise (e.g., paralysis)
* Reading disability/dyslexia
* Prior brain surgery
* Known brain malformation
* Colorblindness
* Heart condition that requires physician approval for physical activity
* Chest pain (with OR without physical activity)
* Loss of balance/dizziness/loss of consciousness
* Bone or joint problem that could be made worse by a change in physical activity
* Medication for blood pressure or a heart condition

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 521 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Bochum Matrices Test | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  BOMAT is a non-verbal, one-dimensional neuropsychological test of Gf. The test consists of a series of 5x3 matrices of patternswith each matrix missing one field. The participant selects one of six possible answers that complete the matrix. The problems range from simple to complex and are all in black-and-white. Participants complete a 15-min practice and have 45 min to complete as many problems as they can (29 total).

SECONDARY OUTCOMES:
Change in Letter Sets | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This test is a measure of Gf. For each problem of the Letter Sets task, the participant is shown 5 sets of letters, with 4 letters in each set. Four of the sets of letters follow a rule, while the fifth set of letters is different from the rest. With the exception of sounds of the sets of letters, shapes of the letters, or potential word formation of the letters, the participant must determine which rule applies to 4 of the letter sets and indicate the 1 letter set that doesn't fit. Participants have 7 minutes to complete as many problems as they can (15 total), with each problem getting progressively more difficult.
Change in Number Series | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This test is a measure of Gf. Participants are shown a series of arithmetic number series and need to select the next number in the series from 5 possible answers at the bottom of the screen. The participant is given 5 practice problems at the beginning of instruction, and must complete as many problems as possible in 5 min (10 total).
Change in Rotation Span | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a test of working memory. Participants must remember a series of arrows presented (16 possible arrows varying in length and direction), while maintaining accuracy on an interleaved letter rotation task (determining if a letter is facing the correct direction after rotation).
Change in Symmetry Span | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a test of working memory. Participants must remember a series of blocks presented (from a 4x4 grid) while maintaining accuracy on an interleaved symmetry judgment task.
Change in Reading Span | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a test of working memory. Participants must remember a series of words presented (18 possible 4-letter words) while maintaining accuracy on an interleaved task where they judge sensible or nonsensical sentences.
Change in Garavan | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  The Garavan task is a serial attention task that measures executive function, specifically task-switching ability. Participants are presented with a series of large and small squares, 10 series/trial in total. Subjects must keep a mental count of how many large and small squares have been presented. For each square, the participant rapidly updates this mental count and then presses the spacebar to see the next square. At the end of the sequence (length is random), a response screen appears and participants report their final count of large and small squares. On a given trial, 11-15 updates are made. Dependent measures are response time for consecutive trials of the same type (no-switch RT) and response time for consecutive trials that differ (switch RT). A cost RT metric can be computed by taking the difference between Switch and No-Switch RT as a measure of set shifting.
Change in Stroop | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  The Stroop task is a measure of executive function, specifically inhibition. In this task, subjects are asked to indicate the color of each word stimulus. The stimulus may be congruent (the word meaning and text color match), or incongruent (the word meaning and text color differ).
Change in Keep Track | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  The Keep Track task measures executive function, specifically updating items held in short-term memory. In the task, a series of word stimuli are presented, each belonging to a category. Subjects must remember only the last item presented from each category.
Change in Immediate and Delayed Free Recall - Words | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a relational memory task. Participants are shown a sequence of 12 words (all 4-letter nouns/verbs), 750 ms for each word. Afterwards, the participant has 30 sec to enter as many words as they can remember from the trial. They do 1 practice trial, followed by 5 test trials. Approximately 20-30 min later, participants are given 90 sec to recall as many words as they can from all 5 previous trials.
Change in Immediate and Delayed Free Recall - Pictures | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a relational memory task. Participants are shown a sequence of 12 images (all objects, no "action" images), 750 ms for each image. Afterwards, the participant has 30 sec to enter words to describe as many images as they recall from the trial (1 word/image). Each image has multiple words that could be accepted as a correct response (i.e., if shown an image of a chimpanzee, answers "chimpanzee" and "monkey" would both be acceptable). They do 1 practice trial of this task, followed by 5 test trials. Approximately 20-30 minutes later, the participant is given 90 sec to recall as many images as they can from all the previous trials.
Change in Paired Associates | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This is a relational memory task. In Paired Associates, a list of 6 unrelated word pairs are presented. At recall, only the first word from each pair is presented. Subjects must enter the second word in the pair. This procedure is repeated with a second list of 6 word pairs. Approximately 20-30 minutes later, the first words from all 12 word pairs are presented. Subjects must enter the second words from each pair.
Change in VO2 Max (relative, percentile) | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Aerobic fitness, defined as maximal oxygen consumption (VO2 max), is assessed using an indirect computerized calorimetry system during a modified Balke treadmill test. During the test, participants' heart rates are monitored using a Polar heart rate monitor, and ratings of perceived exertion are assessed every 2 min. During the test, speed remains constant while incline increases 2-3% every 2 min. Average O2 consumption and respiratory exchange ratio are sampled every 15 sec using a mouthpiece. Relative VO2 max is reported relative to body weight, calculated as ml O2/kg/min. Maximum effort is defined using at least 2 of the following: (1) age-defined maximum heart rate norms (HR > 85% of predicted max HR), (2) respiratory exchange ratio (CO2/O2) >1.1, (3) subjective rate of perceived exertion >17 (of 20), and (4) leveling of VO2 despite increasing aerobic demand. VO2 max percentile is also be reported based on age norms.
Change in Body Mass Index | 2 administrations: within 2 weeks before beginning and after finishing the 16-week intervention period
  BMI is calculated from measures of height and weight
Change in brain structure | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  High-resolution structural MRI scan of brain anatomy using MPRAGE sequence, acquired in sagittal orientation (resolution: 0.9 mm, 192 slices, TR 1900 ms, TE 2.32 ms).
Change in BOLD signal at rest | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Using functional MRI to measure blood-oxygen-level-dependent signal while the subject is at rest and not performing a task
Change in BOLD signal during task | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Functional MRI that measures brain activity (based on hemodynamic response and blood-oxygenation-level dependent signal) during an experimental task.
Change in Object Location Task performance | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Completed during fMRI scanning. In the task, an image with 4 objects is presented on a grid of 9 possible locations. Participants are instructed to memorize the spatial locations of all 4 objects and mentally rotate the grid 90⁰. Participants are then presented with a probe image containing the same 4 objects rotated 90⁰. Participants must indicate whether or not any of the objects changed location in the rotated probe image. There are three possible responses: either all objects match; 1 object moves to a new location; or 2 objects swap locations. This task is a measure of relational memory.
Change in 3-back Task performance | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Completed during fMRI scanning. Participants are presented with a continuous stream of stimuli (either faces or words), and for every stimulus, the participant must indicate (yes/no) whether or not the current stimulus is the same as the one presented three trials back. This task is a measure of working memory.
Change in Diffusion of Water in the brain | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Diffusion tensor imaging (DTI) is a magnetic resonance imaging method that is sensitive to the diffusion of water molecules. Diffusion of water in the brain depends on the tissue type, structural architecture, and presence/absence of barriers within imaging voxels. Using this raw imaging information, diffusion-based properties can be estimated including: 1. fractional anisotropy (FA), which is a measure of whether or not the 3-dimensional diffusion is largely directional (e.g., within an axon; thus, anisotropic diffusion), or if the diffusion is equal in all directions (e.g., within CSF; thus isotropic diffusion); 2. radial diffusivity (RD), which is a measure of how diffusion in the plane transverse to the principal direction of diffusion (i.e., within a cross-section of an axon, rather than down the length of an axon).
Change in single-voxel magnetic resonance spectroscopy (MRS) | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Technique to measure cell metabolites within a single super voxel of the brain (20 mm3), such as N-acetyl aspartate (NAA)
Change in Cerebral Blood Flow | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  During magnetic resonance imaging scans, using the arterial spin labeling technique to acquire multi-slice cerebral blood flow maps
Saliva-based Genetic Biomarkers | One administration, within a week after finishing the 16-week intervention
  Saliva collected from passive drooling, to be analyzed for biomarkers related to fluid intelligence
Height | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Height measured to calculate BMI estimate
Weight | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Weight measured to calculate BMI estimate
Change in Demographics Questionnaire | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Questionnaire that requests age, birth date, sex, race/ethnicity, occupation.
Change in Big Five Inventory (BFI) Questionnaire | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  Personality assessment with five dimensions: openness, conscientiousness, extraversion, agreeableness, and neuroticism
Change in Grit Scale Questionniare | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This questionnaire assesses the personality trait of grit, a characteristic associated with passion and adherence to long-term goals, along with strong motivation to achieve goals despite potential obstacles.
Change in Pittsburgh Sleep Quality Index (PSQI) | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  The PSQI assesses sleep habits on eight dimensions over the past month with 11 open-ended and multiple choice questions. Relevant dimensions include sleep duration, disturbance, latency, day dysfunction, efficiency, quality, use of medications to sleep, and an overall binary score of sleep habits.
Change in Godin-Shepard Leisure Time Physical Activity Questionnaire | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This survey asks about level of physical activity during leisure time in the past month, from which longer-term exercise habits can be extrapolated. By collecting height, weight, and resting heart rate with this measure, a VO2 max estimation can be reliably calculated.
Change in UCLA Loneliness Scale | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This survey asks about the frequency (never, rarely, sometimes, often) of 20 statements regarding feelings of loneliness and social connection.
Change in Need for Cognition | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  This survey asks 45 Likert-type questions regarding the value an individual places upon cognition in daily life.
Change in Implicit Theories of Intelligence Survey (ITIS) | 2 administrations: within a week before beginning and after finishing the 16-week intervention period
  The ITIS asks 8 Likert-type questions regarding personal beliefs about the relative fixedness/malleability of intelligence.
Physical Activity Enjoyment Scale | Administered once, within a week after finishing the 16-week intervention period
  The Physical Activity Enjoyment Scale (PACES) measures individuals' enjoyment with their current activity level.
Post-Experiment Survey | Administered once, within 2 weeks after finishing the 16-week intervention period
  This survey was customized for each arm to assess: participant feedback on the various interventions they experienced; strategies developed and used in cognitive training and active control training; expectancy effects of video game-training, physical fitness training, and mindfulness meditation training; and the contribution of external (outside-study) physical activity/exercise and video game play.
Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q) | Two administrations: within a week before beginning and after finishing the 16-week intervention period
  The Preference and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q) measures individuals' preferences for physical activity type and duration. For instance, does one prefer high-intensity activity for a brief period of time, or low-intensity activity for a longer duration? How does one respond to physical challenge and exhaustion?
Game Feedback - Mind Frontiers | Administered at Sessions 1, 20 (or 24), and 48 of the Mind Frontiers intervention
  Game feedback surveys were developed in-house and administered to evaluate participant responses to cognitive training. These surveys were administered at Sessions 1, 24, and 48 for the 48-session intervention, or at Sessions 1 and 20 for the 20-session intervention. These surveys evaluated enjoyment, engagement, motivation, demand, and frustration with each mini-game.
Game Feedback - Active Control | Administered at Sessions 1, 24, and 48 of Active Control intervention
  Game feedback surveys were developed in-house and administered to evaluate participant responses to active control training. These surveys evaluated enjoyment, engagement, motivation, demand, and frustration with each task.
Army Physical Readiness Test (APRT) | Administered at Session 1 and Session 28 of the fitness intervention
  The APRT is five exercises: (1) 60-yard shuttle run, (2) standing long jump, (3) one-minute of rowers, (4) one-minute of push-ups, and (5) a 1.5 mile run
Heart rate | Data collected continuously during at all 28 fitness intervention sessions
  Participants' heart rates were monitored using Polar heart rate monitor E600 during all sessions of the fitness intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aron K Barbey, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign; Arthur F Kramer, Ph.D., Principal Investigator — Northeastern University; Neal J Cohen, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign; Charles H Hillman, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Aggregate data will be shared. Details of individual participant data to be shared are still under discussion.

REFERENCES:
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Colcombe SJ, Kramer AF, Erickson KI, Scalf P, McAuley E, Cohen NJ, Webb A, Jerome GJ, Marquez DX, Elavsky S. Cardiovascular fitness, cortical plasticity, and aging. Proc Natl Acad Sci U S A. 2004 Mar 2;101(9):3316-21. doi: 10.1073/pnas.0400266101. Epub 2004 Feb 20. PMID 14978288
- [Background] Chaddock L, Erickson KI, Prakash RS, VanPatter M, Voss MW, Pontifex MB, Raine LB, Hillman CH, Kramer AF. Basal ganglia volume is associated with aerobic fitness in preadolescent children. Dev Neurosci. 2010 Aug;32(3):249-56. doi: 10.1159/000316648. Epub 2010 Aug 6. PMID 20693803
- [Background] Blackwell LS, Trzesniewski KH, Dweck CS. Implicit theories of intelligence predict achievement across an adolescent transition: a longitudinal study and an intervention. Child Dev. 2007 Jan-Feb;78(1):246-63. doi: 10.1111/j.1467-8624.2007.00995.x. PMID 17328703
- [Background] Hillman CH, Kramer AF, Belopolsky AV, Smith DP. A cross-sectional examination of age and physical activity on performance and event-related brain potentials in a task switching paradigm. Int J Psychophysiol. 2006 Jan;59(1):30-9. doi: 10.1016/j.ijpsycho.2005.04.009. PMID 16413382
- [Background] Kamijo K, O'Leary KC, Pontifex MB, Themanson JR, Hillman CH. The relation of aerobic fitness to neuroelectric indices of cognitive and motor task preparation. Psychophysiology. 2010 Sep;47(5):814-21. doi: 10.1111/j.1469-8986.2010.00992.x. Epub 2010 Mar 23. PMID 20345598
- [Background] Liu-Ambrose T, Nagamatsu LS, Graf P, Beattie BL, Ashe MC, Handy TC. Resistance training and executive functions: a 12-month randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):170-8. doi: 10.1001/archinternmed.2009.494. PMID 20101012
- [Background] Monti JM, Hillman CH, Cohen NJ. Aerobic fitness enhances relational memory in preadolescent children: the FITKids randomized control trial. Hippocampus. 2012 Sep;22(9):1876-82. doi: 10.1002/hipo.22023. Epub 2012 Apr 23. PMID 22522428
- [Background] Pontifex MB, Hillman CH, Polich J. Age, physical fitness, and attention: P3a and P3b. Psychophysiology. 2009 Mar;46(2):379-87. doi: 10.1111/j.1469-8986.2008.00782.x. Epub 2009 Jan 26. PMID 19170947
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924
- [Background] Themanson JR, Hillman CH, Curtin JJ. Age and physical activity influences on action monitoring during task switching. Neurobiol Aging. 2006 Sep;27(9):1335-45. doi: 10.1016/j.neurobiolaging.2005.07.002. Epub 2005 Aug 15. PMID 16102874
- [Background] Themanson JR, Pontifex MB, Hillman CH. Fitness and action monitoring: evidence for improved cognitive flexibility in young adults. Neuroscience. 2008 Nov 19;157(2):319-28. doi: 10.1016/j.neuroscience.2008.09.014. Epub 2008 Sep 13. PMID 18845227
- [Background] Voss MW, Erickson KI, Prakash RS, Chaddock L, Malkowski E, Alves H, Kim JS, Morris KS, White SM, Wojcicki TR, Hu L, Szabo A, Klamm E, McAuley E, Kramer AF. Functional connectivity: a source of variance in the association between cardiorespiratory fitness and cognition? Neuropsychologia. 2010 Apr;48(5):1394-406. doi: 10.1016/j.neuropsychologia.2010.01.005. Epub 2010 Jan 15. PMID 20079755
- [Background] Voss MW, Heo S, Prakash RS, Erickson KI, Alves H, Chaddock L, Szabo AN, Mailey EL, Wojcicki TR, White SM, Gothe N, McAuley E, Sutton BP, Kramer AF. The influence of aerobic fitness on cerebral white matter integrity and cognitive function in older adults: results of a one-year exercise intervention. Hum Brain Mapp. 2013 Nov;34(11):2972-85. doi: 10.1002/hbm.22119. Epub 2012 Jun 5. PMID 22674729
- [Background] Weinstein AM, Voss MW, Prakash RS, Chaddock L, Szabo A, White SM, Wojcicki TR, Mailey E, McAuley E, Kramer AF, Erickson KI. The association between aerobic fitness and executive function is mediated by prefrontal cortex volume. Brain Behav Immun. 2012 Jul;26(5):811-9. doi: 10.1016/j.bbi.2011.11.008. Epub 2011 Dec 7. PMID 22172477
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Ball K, Edwards JD, Ross LA. The impact of speed of processing training on cognitive and everyday functions. J Gerontol B Psychol Sci Soc Sci. 2007 Jun;62 Spec No 1:19-31. doi: 10.1093/geronb/62.special_issue_1.19. PMID 17565162
- [Background] Baniqued PL, Lee H, Voss MW, Basak C, Cosman JD, Desouza S, Severson J, Salthouse TA, Kramer AF. Selling points: What cognitive abilities are tapped by casual video games? Acta Psychol (Amst). 2013 Jan;142(1):74-86. doi: 10.1016/j.actpsy.2012.11.009. Epub 2012 Dec 17. PMID 23246789
- [Background] Dahlin E, Neely AS, Larsson A, Backman L, Nyberg L. Transfer of learning after updating training mediated by the striatum. Science. 2008 Jun 13;320(5882):1510-2. doi: 10.1126/science.1155466. PMID 18556560
- [Background] Olesen PJ, Westerberg H, Klingberg T. Increased prefrontal and parietal activity after training of working memory. Nat Neurosci. 2004 Jan;7(1):75-9. doi: 10.1038/nn1165. Epub 2003 Dec 14. PMID 14699419
- [Background] Zook NA, Davalos DB, Delosh EL, Davis HP. Working memory, inhibition, and fluid intelligence as predictors of performance on Tower of Hanoi and London tasks. Brain Cogn. 2004 Dec;56(3):286-92. doi: 10.1016/j.bandc.2004.07.003. PMID 15522766
- [Background] Mackey AP, Hill SS, Stone SI, Bunge SA. Differential effects of reasoning and speed training in children. Dev Sci. 2011 May;14(3):582-90. doi: 10.1111/j.1467-7687.2010.01005.x. Epub 2010 Nov 23. PMID 21477196
- [Background] Karbach J, Kray J. How useful is executive control training? Age differences in near and far transfer of task-switching training. Dev Sci. 2009 Nov;12(6):978-90. doi: 10.1111/j.1467-7687.2009.00846.x. PMID 19840052
- [Background] Barbey AK, Colom R, Grafman J. Distributed neural system for emotional intelligence revealed by lesion mapping. Soc Cogn Affect Neurosci. 2014 Mar;9(3):265-72. doi: 10.1093/scan/nss124. Epub 2012 Nov 19. PMID 23171618
- [Background] Chaddock L, Erickson KI, Prakash RS, Kim JS, Voss MW, Vanpatter M, Pontifex MB, Raine LB, Konkel A, Hillman CH, Cohen NJ, Kramer AF. A neuroimaging investigation of the association between aerobic fitness, hippocampal volume, and memory performance in preadolescent children. Brain Res. 2010 Oct 28;1358:172-83. doi: 10.1016/j.brainres.2010.08.049. Epub 2010 Aug 22. PMID 20735996
- [Background] Antal A, Nitsche MA, Kincses TZ, Kruse W, Hoffmann KP, Paulus W. Facilitation of visuo-motor learning by transcranial direct current stimulation of the motor and extrastriate visual areas in humans. Eur J Neurosci. 2004 May;19(10):2888-92. doi: 10.1111/j.1460-9568.2004.03367.x. PMID 15147322
- [Background] Boggio PS, Fregni F, Valasek C, Ellwood S, Chi R, Gallate J, Pascual-Leone A, Snyder A. Temporal lobe cortical electrical stimulation during the encoding and retrieval phase reduces false memories. PLoS One. 2009;4(3):e4959. doi: 10.1371/journal.pone.0004959. Epub 2009 Mar 25. PMID 19319182
- [Background] Coffman BA, Trumbo MC, Clark VP. Enhancement of object detection with transcranial direct current stimulation is associated with increased attention. BMC Neurosci. 2012 Sep 10;13:108. doi: 10.1186/1471-2202-13-108. PMID 22963503
- [Background] Utz KS, Dimova V, Oppenlander K, Kerkhoff G. Electrified minds: transcranial direct current stimulation (tDCS) and galvanic vestibular stimulation (GVS) as methods of non-invasive brain stimulation in neuropsychology--a review of current data and future implications. Neuropsychologia. 2010 Aug;48(10):2789-810. doi: 10.1016/j.neuropsychologia.2010.06.002. Epub 2010 Jun 11. PMID 20542047
- [Background] Coffman BA, Trumbo MC, Flores RA, Garcia CM, van der Merwe AJ, Wassermann EM, Weisend MP, Clark VP. Impact of tDCS on performance and learning of target detection: interaction with stimulus characteristics and experimental design. Neuropsychologia. 2012 Jun;50(7):1594-602. doi: 10.1016/j.neuropsychologia.2012.03.012. Epub 2012 Mar 19. PMID 22450198
- [Background] Clark VP, Coffman BA, Mayer AR, Weisend MP, Lane TD, Calhoun VD, Raybourn EM, Garcia CM, Wassermann EM. TDCS guided using fMRI significantly accelerates learning to identify concealed objects. Neuroimage. 2012 Jan 2;59(1):117-28. doi: 10.1016/j.neuroimage.2010.11.036. Epub 2010 Nov 19. PMID 21094258
- [Background] Ditye T, Jacobson L, Walsh V, Lavidor M. Modulating behavioral inhibition by tDCS combined with cognitive training. Exp Brain Res. 2012 Jun;219(3):363-8. doi: 10.1007/s00221-012-3098-4. Epub 2012 Apr 25. PMID 22532165
- [Background] Reis J, Schambra HM, Cohen LG, Buch ER, Fritsch B, Zarahn E, Celnik PA, Krakauer JW. Noninvasive cortical stimulation enhances motor skill acquisition over multiple days through an effect on consolidation. Proc Natl Acad Sci U S A. 2009 Feb 3;106(5):1590-5. doi: 10.1073/pnas.0805413106. Epub 2009 Jan 21. PMID 19164589
- [Background] Redick TS, Shipstead Z, Harrison TL, Hicks KL, Fried DE, Hambrick DZ, Kane MJ, Engle RW. No evidence of intelligence improvement after working memory training: a randomized, placebo-controlled study. J Exp Psychol Gen. 2013 May;142(2):359-79. doi: 10.1037/a0029082. Epub 2012 Jun 18. PMID 22708717
- [Background] Gaspar JG, Neider MB, Simons DJ, McCarley JS, Kramer AF. Change detection: training and transfer. PLoS One. 2013 Jun 28;8(6):e67781. doi: 10.1371/journal.pone.0067781. Print 2013. PMID 23840775
- [Background] Baniqued PL, Allen CM, Kranz MB, Johnson K, Sipolins A, Dickens C, Ward N, Geyer A, Kramer AF. Working Memory, Reasoning, and Task Switching Training: Transfer Effects, Limitations, and Great Expectations? PLoS One. 2015 Nov 10;10(11):e0142169. doi: 10.1371/journal.pone.0142169. eCollection 2015. PMID 26555341
- [Background] Shallice T. Specific impairments of planning. Philos Trans R Soc Lond B Biol Sci. 1982 Jun 25;298(1089):199-209. doi: 10.1098/rstb.1982.0082. PMID 6125971
- [Background] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Shah P, Miyake A. The separability of working memory resources for spatial thinking and language processing: an individual differences approach. J Exp Psychol Gen. 1996 Mar;125(1):4-27. doi: 10.1037//0096-3445.125.1.4. PMID 8851737
- [Background] Unsworth N, Redick TS, Heitz RP, Broadway JM, Engle RW. Complex working memory span tasks and higher-order cognition: a latent-variable analysis of the relationship between processing and storage. Memory. 2009 Aug;17(6):635-54. doi: 10.1080/09658210902998047. Epub 2009 Jun 17. PMID 19536691
- [Background] Engle RW, Tuholski SW, Laughlin JE, Conway ARA. Working memory, short-term memory, and general fluid intelligence: a latent-variable approach. J Exp Psychol Gen. 1999 Sep;128(3):309-331. doi: 10.1037//0096-3445.128.3.309. PMID 10513398
- [Background] Garavan H. Serial attention within working memory. Mem Cognit. 1998 Mar;26(2):263-76. doi: 10.3758/bf03201138. PMID 9584434
- [Background] YNTEMA DB. Keeping track of several things at once. Hum Factors. 1963 Feb;5:7-17. doi: 10.1177/001872086300500102. No abstract available. PMID 14002586
- [Background] Unsworth N, Spillers GJ, Brewer GA. The contributions of primary and secondary memory to working memory capacity: an individual differences analysis of immediate free recall. J Exp Psychol Learn Mem Cogn. 2010 Jan;36(1):240-7. doi: 10.1037/a0017739. PMID 20053060
- [Background] Auerbach EJ, Xu J, Yacoub E, Moeller S, Ugurbil K. Multiband accelerated spin-echo echo planar imaging with reduced peak RF power using time-shifted RF pulses. Magn Reson Med. 2013 May;69(5):1261-7. doi: 10.1002/mrm.24719. Epub 2013 Mar 6. PMID 23468087
- [Background] Ouyang C, Sutton BP. Pseudo-continuous transfer insensitive labeling technique. Magn Reson Med. 2011 Sep;66(3):768-76. doi: 10.1002/mrm.22815. Epub 2011 Mar 4. PMID 21381103
- [Background] Gray JR, Chabris CF, Braver TS. Neural mechanisms of general fluid intelligence. Nat Neurosci. 2003 Mar;6(3):316-22. doi: 10.1038/nn1014. PMID 12592404
- [Background] Hannula DE, Ranganath C. Medial temporal lobe activity predicts successful relational memory binding. J Neurosci. 2008 Jan 2;28(1):116-24. doi: 10.1523/JNEUROSCI.3086-07.2008. PMID 18171929
- [Background] Soares JM, Marques P, Alves V, Sousa N. A hitchhiker's guide to diffusion tensor imaging. Front Neurosci. 2013 Mar 12;7:31. doi: 10.3389/fnins.2013.00031. eCollection 2013. PMID 23486659
- [Background] Duckworth AL, Peterson C, Matthews MD, Kelly DR. Grit: perseverance and passion for long-term goals. J Pers Soc Psychol. 2007 Jun;92(6):1087-101. doi: 10.1037/0022-3514.92.6.1087. PMID 17547490
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Hossip, R, Turck, D, Hasella, A. Bocumer Matrizentest: BOMAT-Advanced-Short Version. Göttingen: Hogrefe Ltd; 1999.
- [Background] Moody, DE. Can intelligence be increased by training on a task of working memory? Intelligence. 2009; 37(4):327-328.
- [Background] French, JW, Harmann, HH, Dermen, D. Manual for kit of factor-referenced cognitive tests. New Jersey: Educational Testing Service; 1976. p. 109-113
- [Background] Bernreuter, RG, Goodman, CH. A study of the Thurstone Primary Mental Abilities Tests applied to freshman engineering students. J Exp Psychol Gen. 1941; 32(1):55-60.
- [Background] Stroop, JR. Studies of inference in serial verbal reactions. J Exp Psychol. 1935;18(6):643-662.
- [Background] American College of Sports Medicine. ACSM's guidelines for exercise testing and prescription. Philadelphia, PA: Wolters Kluwer/Lippincott Williams & Wilkins; 2010.
- [Background] John, O, Donahue, EM, Kentle, RL. The Big Five Inventory - Versions 4a and 54. Berkeley, CA: University of California Institute of Personality and Social Research; 1991.
- [Background] Cacioppo, JT, Petty, RE. The need for cognition. J Pers Soc Psychol. 1982; 42(1): 116.
- [Background] Kendzierski, D, DeCarlo, KJ. Physical Activity Enjoyment Scale: Two validation studies. J Sport Exerc Psych. 1991; 13(1): 50-64.
- [Background] Ekkekakis, P, Hall, E, Petruzello, SJ. Some like it vigorous: Measuring individual differences in the preference for and tolerance of exercise intensity. J Sport Exerc Psych. 2005; 27, 350-374.
- [Result] Watson PD, Paul EJ, Cooke GE, Ward N, Monti JM, Horecka KM, Allen CM, Hillman CH, Cohen NJ, Kramer AF, Barbey AK. Underlying sources of cognitive-anatomical variation in multi-modal neuroimaging and cognitive testing. Neuroimage. 2016 Apr 1;129:439-449. doi: 10.1016/j.neuroimage.2016.01.023. Epub 2016 Jan 22. PMID 26808332
- [Result] Greenlee, T, Greene, DR, Ward, NJ, Reeser, GE, Allen, CM, Baumgartner, NW, Cohen, NJ, Kramer, AF, Barbey, AK, Hillman, CH. Effectiveness of a 16-Week High Intensity Cardio-Resistance Training (HICRT) Program in young and middle aged adults. Poster session presented at: American College of Sports Medicine 2016 Conference; 2016 Jun 3; Boston, MA.
- [Result] Baumgartner, NW, Covello, AR, Reeser, GE, Cohen, NJ, Kramer, AF, Barbey, AK, Hillman, CH, Khan, NA. Moderate to vigorous physical activity influences aerobic capacity independent of body composition. Poster session presented at: American College of Sports Medicine 2016 Conference; 2016 Jun; Boston, MA.
- [Result] Covello, A, Baumgartner, NW, Curran, MR, Reeser, GE, Cohen, NJ, Kramer, AF, Hillman, CH, Barbey, AK, Khan, NA. The sexual dimorphic relationship between dietary fiber intake and visceral adipose tissue. Abstract accepted to: Experimental Biology 2016 Meeting; 2016 Apr; San Diego, CA.